CLINICAL TRIAL: NCT01322828
Title: Randomized Control Trial Comparing Single Incision Versus Double Incision Surgery to Repair Distal Bicep Tendon Ruptures
Brief Title: Trial Comparing Single Versus Double Incision to Repair Distal Bicep Tendon Ruptures
Acronym: BRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hand and Upper Limb Clinic, Canada (Network)
Responsible Party: Dr. Joy MacDermid, Hand and Upper Limb Centre, St. Josephs Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HULCbicep
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Distal Bicep Tendon Rupture
Keywords: Bicep; Tendon; Distal; Ruptures; Randomized; Surgery
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single incision repair of distal bicep tendon rupture (Active Comparator): In this treatment arm patients will have a single incision technique used to repair their distal bicep tendon rupture
  Interventions: Procedure: Distal bicep tendon reconstruction
- Double incision repair of distal bicep tendon rupture (Active Comparator): In this treatment arm, patients will have a double incision technique used to repair their distal bicep tendon rupture.
  Interventions: Procedure: Distal bicep tendon reconstruction

INTERVENTIONS:
Procedure: Distal bicep tendon reconstruction — Randomized to either a single incision technique or a double incision technique.

SUMMARY:
The purpose of this study to to determine whether a single incision technique or a double incision technique is more effective in the surgical treatment of distal bicep tendon ruptures. Patients will be randomized to one of the two techniques upon consenting to the study. Prior to surgery patients will have their elbow flexion, extension, pronation, and supination strength measured. Elbow Range of motion will also be measured in each of these four movements. A number of subjective questionnaires will also be administered to the patient prior to surgery. The identical objective tests and subjective questionnaires will be completed by the patient at intervals of three months, six months, one year, and two years following their surgery. Additional information from patients clinical visits may also be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Complete rupture of the Distal Bicep tendon
* Acute bicep tendon rupture (< 10 days since rupture)
* 18 years of age and older

Exclusion Criteria:

* Partial rupture of the Distal Bicep tendon
* Chronic bicep tendon Ruptures (>10 days since rupture)
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDermid, MSc, PhD, Principal Investigator — Hand and Upper Limb Centre, St Joseph's health Care
Locations (2):
- Canada (2):
  - Hand and Upper Limb Centre, St. Joseph's Health Care, London, Ontario
  - Hand and Upper Limb Centre, London, Ontario